CLINICAL TRIAL: NCT01447316
Title: Impact of Bariatric Surgery on Short Term Weight Loss- Related Changes in Gait and Quality of Life
Brief Title: Bariatric Surgery on Short Term Weight Loss- Related Changes in Gait
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 332-2009
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Obesity, Morbid
Keywords: body composition; gait; quality of life; Patients; undergoing; bariatric surgery.
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric surgery: Patients undergoing bariatric surgery for weight loss.
  Interventions: Other: Subject outcomes following bariatric surgery

INTERVENTIONS:
Other: Subject outcomes following bariatric surgery — Subject outcomes (body composition, gait analysis, lower extremity joint pain and perceived quality of life) measured at per-op, 2, 4 weeks and 3 months.

SUMMARY:
This is a short term study of the effects of bariatric surgery on body composition, gait parameters during walking, lower extremity joint pain and quality of life (QOL) in morbidly obese patients who are already scheduled for a bariatric surgical procedure.

DETAILED DESCRIPTION:
This is a prospective, exploratory, short term study of the effects of bariatric surgery on body composition, gait parameters during walking, lower extremity joint pain and quality of life (QOL) in morbidly obese patients. All patients who enroll have already agreed to undergo the bariatric procedure with their respective surgeon; the study team will simply follow specific outcome measures in addition to their normal clinical care at two time points after the surgery (week 4 and month 3).

ELIGIBILITY:
Inclusion Criteria:

* no urgent need for bariatric procedure
* 21-65 years of age
* body mass index (BMI) 35 kg/m2 or greater, defined as morbid obesity
* waist circumference of < 66 inches
* able to walk independently

Exclusion Criteria:

* < 21 or > 65 years of age
* pregnancy; psychiatric conditions; binge eating patterns; Prader-Willi syndrome; drug dependency; dementia or other neurodegenerative diseases that would preclude appropriate cognitive or physical ability to perform study protocol
* uncontrolled diabetes (not using meds)
* waist circumference of > 66 inches
* orthopedic conditions that prevent ambulation (severe painful osteoarthritis of the hip or knee)
* patient is wheelchair bound

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will be patients already scheduled to undergo bariatric surgery for weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Body Composition, describes change in body composition from pre-op levels | Describes change over a period of 4 weeks; measured at pre-op, 2 and 4 weeks following surgery
  To track changes in body composition and mass during the study, body weight body fat mass, fat free mass will be collected prior to and 2 and 4 weeks after the bariatric surgery using air plethysmography. Air plethysmography (using the BOD POD®) is a reliable technique of body volume and composition, and has been validated for use in obese individuals and is highly correlated to the gold standard of body composition assessment, underwater weighing.

SECONDARY OUTCOMES:
Gait Analysis, describes change in gait parameters from pre-op levels | Describes changes in gait parameters over a 3 month period; measured at pre-op, 4 weeks and 3 months following surgery.
  The gait analysis involves walking on a 26' long portable gait mat (GaitRite®). The mat is a cushioned thin mat filled with pressure sensors. Participants will be asked to walk at a self-selected, comfortable pace across the 26 foot long mat. This normal self-selected pace will be performed three times and the values will be averaged for the three trials. The participant will then be asked to walk as quickly as possible across the mat and the velocity to reach 20' will be determined. This will be repeated two more times for a total of 3 trials.
Lower Extremity Joint Pain, describes change from pre-op using a Visual Analog Scale (VAS). | Describes change in lower extremity joint pain over a period of 3 months; measured with a (VAS) at per-op, 4 weeks and 3 months following surgery
  Joint pain intensity will be self-assessed by a 10 cm (VAS) with terminal descriptors (anchors of 0 cm = no pain; 10 cm = worst possible pain). The (VAS) is an accepted outcome measure for chronic pain.
Medical Outcomes Short Form (SF-36), describes change in perceived quality of life (QOL) | Describes perceived (QOL) over a period of 3 months, measured at pre-op, 4 weeks and 3 months following surgery
  The (SF36) is an instrument that assesses overall health-related (QOL). The (SF36) is comprised of eight subscales, each ranging from 0-100 points, with higher scores representing better health. The (SF36) has been recommended for use following bariatric surgery to capture meaningful changes in (QOL).

CONTACTS AND LOCATIONS:
Overall Officials: Heather K Vincent, Ph.D., Principal Investigator — University of Florida Department of Orthopaedics and Rehabilitation
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States